CLINICAL TRIAL: NCT00282425
Title: Non-myeloablative Allogeneic Hematopoietic Stem Cell Transplantation (NST) for Patients With Systemic Sclerosis
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation (NST) for Patients With Systemic Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No subject enrolled since 2009
Sponsor: Richard Burt, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Burt, MD, MD, Northwestern University
Organization: Northwestern University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD Scl.Allo2005
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Hematopoietic stem cell transplantation (Experimental): Allogeneic Hematopoietic stem cell transplantation will be performed on eligible patients
  Interventions: Biological: Hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: Hematopoietic stem cell transplantation — Allogeneic Hematopoietic stem cell transplantation

SUMMARY:
Scleroderma is disease believed to be due to immune cells, cells which normally protect the body but are now causing damage to the body. There has not been any treatment that has been effective in treating this disease. The likelihood of progression of the disease to severe disability and death is high. This study is designed to examine whether treating patients with high dose Cyclophosphamide and Fludarabine (drugs which reduce the function of your immune system) and CAMPATH-1H (a protein that kills the immune cells that are thought to be causing the disease), followed by return of blood stem cells that have been previously collected from patients brother or sister will stop or reverse the disease. The purpose of the Cyclophosphamide, Fludarabine and CAMPATH-1H is to decrease immune system. The purpose of the stem cell infusion is to restore blood production, which will be severely impaired by the Cyclophosphamide, Fludarabine and CAMPATH-1H, and to produce a normal immune system that will no longer attack the body.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Age 18 to 55 years old
2. An established diagnosis of scleroderma (84)
3. Diffuse cutaneous scleroderma with involvement proximal to the elbow or knee and a Rodnan score (see Appendix III) of > 14 (85)

And one of the following:

1. DLCO < 80% of predicted or decrease in lung function (TLC, DLCO or FEV1) of 10% or more over 12 months
2. Active alveolitis on bronchoalveolar lavage
3. Pulmonary fibrosis or alveolitis on CT scan or CXR
4. Elevated ESR greater than or equal to 25mm/hour confirmed on a second occasion at least two weeks apart without evidence of active infectious process.
5. Abnormal EKG (low QRS voltage, or ventricular hypertrophy) or left ventricle (LV) diastolic dysfunction (expressed by an inverted E/A ratio which represents early and late filling of the LV during atrial contraction) or LV wall thickness
6. Since pulmonary disease independent of skin score (NEJM, 2006, 345:25 2655-2709) carries a poor prognosis, patient may be enroled for only lung involvement defined as active alveolitis on BAL or ground-glass opacity on CT, a DLCO < 80% predicted or decrease in lung function (TLC), DLCO, FVC) of 10% or more in last 12 months.

Patient Exclusion Criteria:

1. Poor performance status (ECOG > or =2) at the time of entry, unless due to disease.
2. Significant end organ damage such as:

   1. LVEF <40% or deterioration of LVEF during exercise test on MUGA or echocardiogram
   2. Untreated life-threatening arrhythmia
   3. Active ischemic heart disease or heart failure
   4. DLCO less than 45% of predicted value, unless due to disease.
   5. Pulmonary hypertension (estimated systolic pulmonary arterial pressure >40 mmHg by Doppler echocardiography or measurement by pulmonary arterial catheter)
   6. Serum creatinine > 2.0 mg/dl
   7. Liver cirrhosis, transaminases >3x of normal limits or bilirubin >2.0 unless due to Gilberts disease
3. HIV positive
4. Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment
5. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.
6. Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy
7. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
8. Inability to give informed consent
9. Age <18 or > 55 years old

Donor Inclusion Criteria:

1. Donor must be a HLA identical sibling or HLA matched cord blood donor
2. If donor is HLA matched sibling, donor must be > 18 years of age and less than 50 years old
3. If multiple HLA matched donors are available, preference will be given to same sex, same CMV status, or in the case of cord blood higher nucleated cell count
4. If donor is HLA matched cord blood, cord blood stem cells will be obtained from the New York Blood Center Cord Blood Registry (Tel 212-570-3230) which is an internationally recognized registry or, if a match is not available, from Stemcyte (626-821-9860) which is a commercial registry that specializes in minority donors. One unit of HLA matched cord blood unit will be infused on day zero

Donor Exclusion Criteria:

1. Age > 50 years old or <18 years old
2. HIV positive
3. Active ischemic heart disease or heart failure
4. Acute or chronic active hepatitis
5. Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the donor to tolerate stem cell collection
6. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.
7. Positive pregnancy test
8. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
9. Major hematological abnormalities such as platelet count less than 100,000/ul, ANC less than 1000/ul
10. If donor is sibling must collect a minimum of 2. 106CD34+ cells/kg to proceed to transplant
11. If donor is cord blood unit(s) then a minimum number of nucleated cells available must be more than 2 x 107 /kg. To achieve this number of nucleated cells, two units of HLA matched cord blood may be utilized. (Wagner JE Blood. 2005 Feb 1;105(3):1343-7)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Survival; Disease improvement;Time to disease progression | 5 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States